CLINICAL TRIAL: NCT07385040
Title: Comparison of Intravenous Lignocain and Intravenous Dexmedetomidine for Attenuation of Hemodynamic Stress Response to Direct Laryngoscopy and Endotracheal Intubation
Brief Title: Comparison of IV Lignocain and IV Dexmedetomidine for Attenuation of Laryngoscopic Stress Response to Direct Laryngoscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, Dr. Maryam, Consultant Anesthesiologist, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERC-000072/SMBBIT/Aproval/2023
Record Dates: First submitted 2025-12-07; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Tachycardia; Hypertension; Mean Arterial Pressure
Keywords: Direct laryngoscopy; Hemodynamic stress response; Lignocaine; Dexmedetomidine
MeSH Terms: conditions — Tachycardia; Hypertension

STUDY DESIGN:
Intervention Model Description: Single blinded, randomised control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Active Comparator): Group L received IV Lignocain 1.5mg/kg before induction.
  Interventions: Drug: Intravenous Lignocain
- Group D (Active Comparator): Group D received IV Dexmedetomidine infusion 10mics/ kg over 10min before induction
  Interventions: Drug: Intravenous Dexmedetomidine infusion

INTERVENTIONS:
Drug: Intravenous Dexmedetomidine infusion — Dexmedetomidine infusion with dose of 10mics/kg given 10min before induction
  Arms: Group D
Drug: Intravenous Lignocain — Intravenous ligoncain 1.5mg/kg given 90sec before induction.
  Arms: Group L

SUMMARY:
Hemodymanic stress response to direct laryngoscopy and endotracheal intubation is a known phenomenon that occur in almost every patient undergoing general anesthesia before surgical procedure. This response leads to sudden rise in heart rate and blood pressure which may cause serious complications in compromised patients having cardiovascular diseases. There are certain drugs which are used to blunt this response and to prevent the life threatening complications. Intravenous Lignocain is commonly used drug to blunt the laryngoscopic response in our setup. Intravenous Dexmedetomidine is a newer and rarely used drug to prevent stress response to direct laryngoscopy and endotracheal intubation. This study aims to compare the efficacy of both the drugs to provide better control of complications like Arrythmias, stroke and cardiovascular instability.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing general anesthesia for any elective surgery Having ASA 1 or 2 Having mallapatti 1 or 2 Having BMI in between 18-30 kg/m2

Exclusion Criteria:

Lack of consent Anticipated difficult airway Pregnancy Sensitivity to either drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic stress response | 1 minute and 3 minute after endotracheal intubation
  Rise in Heart rate and mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Maryam, Principal Investigator — Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Locations (1):
- Maryam, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahiswar AP, Dubey PK, Ranjan A. Comparison between dexmedetomidine and fentanyl bolus in attenuating the stress response to laryngoscopy and tracheal intubation: a randomized double-blind trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):103-109. doi: 10.1016/j.bjane.2021.02.060. Epub 2021 May 14. PMID: 34000325; PMCID: PMC9373229.
- See also: J NTR Univ Health Sci 2015;4:86-90 — https://www.researchgate.net/publication/279221880_Comparison_of_intravenous_lignocaine_and_intravenous_dexmedetomidine_for_attenuation_of_hemodynamic_stress_response_to_laryngoscopy_and_endotracheal_intubation